CLINICAL TRIAL: NCT04087226
Title: Comparative Evaluation of Gingival Displacement by Polytetrafluoroethylene (PTFE) & Conventional Retraction Cord- A Randomized Control Trial
Brief Title: Gingival Displacement by Polytetrafluoroethylene & Conventional Retraction Cord
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Humera Nasim, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 54321
Record Dates: First submitted 2019-09-04; First posted 2019-09-12 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Gingival Pocket
Keywords: Polytetrafluoroethylene; Retraction; Soft tissue Management; Retraction cord
MeSH Terms: conditions — Gingival Pocket

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Retraction Cord (Active Comparator)
  Interventions: Device: PTFE Retraction Cord
- PTFE Retraction Cord (Experimental)
  Interventions: Device: PTFE Retraction Cord

INTERVENTIONS:
Device: PTFE Retraction Cord — Polytetrafluoroethylene (PTFE) Retraction cord will be gently applied in gingival sulcus with minimal pressure. The intervention will be applied for three minutes in gingival sulcus, followed by a two stage addition silicone impression.

SUMMARY:
To achieve harmony between restoration and surrounding periodontium, soft tissue management plays a pivotal role. Various Gingival displacement techniques show varying results in achieving the goals of displacement. The most preferred method of displacement by dental practitioners is through conventional retraction cord made up of cotton, which besides its advantages, poses certain drawbacks, including low tear strength, high friction, and fiber remnants within the sulcus.

Polytetrafluoroethylene (PTFE) retraction cord, is a fluoropolymer, known for its high tear strength, low friction, and bio-compatibility.

This study aims to determine the difference of horizontal gingival displacement between PTFE and conventional retraction cord.

Participants inducted in this study will be assessed for eligibility. qualifying subjects will receive crown preparation for Porcelain-fused to-metal crown. subjects will then be randomly allocated to either of the two arms of intervention. After making a pre-displacement impression, Retraction cord will be applied for 3 minutes, then removed to record post-displacement impression.

the difference in pre and post-displacement mean gingival sulcus width will be assessed by a stereomicroscope using image analysis software.

ELIGIBILITY:
Inclusion Criteria:

* Indication of full veneer crown

  * Age group: 18-60 years
  * Probing Depth 2-3mm and no bleeding on probing
  * No signs of gingival/periodontal disease

Exclusion Criteria:

* Indication of subgingival margin location

  * Developmental anomaly (anatomical) affecting abutment tooth
  * Bleeding disorder
  * Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Difference between Mean Horizontal Gingival Displacement by PTFE retraction cord and Conventional retraction cord among sixty participants as assessed by Stereomicroscope. | 3 minutes after displacement

SECONDARY OUTCOMES:
Difference between Post-displacement Bleeding by PTFE and conventional retraction cord among sixty participants by visual assessment | immediately after cord removal
Difference between ease of Application of PTFE and conventional retraction cord among sixty participants. | immediately after cord removal

CONTACTS AND LOCATIONS:
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan